CLINICAL TRIAL: NCT03852147
Title: Individualized Hemodynamic Optimization by Indirect Measurement of the Respiratory Quotient in Major Surgery: Prospective Randomized Multicentre Open-Label Study (OPHIQUE) Individualized Optimization by Indirect Measurement of the Respiratory Quotient
Acronym: OPHIQUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: st isabelle health center, abbeville (Unknown); Centre Hospitalier Universitaire de Caen (Other); Centre Hospitalier VALENCIENNES (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2018_843_0014
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Post-Op Complication; Respiratory Complication
Keywords: respiratory quotient; post operative complications; anaerobic metabolism
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): hemodynamic management of patients is done according to usual practices by maintenance of blood pressure by norepinephrine as well as optimization of SV by vascular filling and use of dobutamine if necessary.
  Interventions: Procedure: : hemodynamic management
- Experimental group (Experimental): perioperative hemodynamic management is based on an algorithm that includes RQ measurement and includes volume expansion, norepinephrine, FiO2 enhancement, RBC transfusion and dobutamine.
  Interventions: Procedure: : hemodynamic management

INTERVENTIONS:
Procedure: : hemodynamic management — Control group: hemodynamic management of patients is done according to usual practices by maintenance of blood pressure by norepinephrine as well as optimization of SV by vascular filling and use of dobutamine if necessary.
  Experimental group: perioperative hemodynamic management is based on an algorithm that includes RQ measurement and includes volume expansion, norepinephrine, FiO2 enhancement, RBC transfusion and dobutamine.

SUMMARY:
The measurement of the inspired / expired fractions in O2 and CO2 is part of the daily monitoring of the intubated-ventilated patient in the operating theater. The ratio of VCO2 to VO2 (respiratory quotient (RQ)) is a non-invasive indirect measure of anaerobic metabolism of the patient, and an indirect reflection of tissue perfusion. We hypothesize that a hemodynamic optimization in major surgery individualized by non-invasive continuous measurement of the RQ would optimize TaO2 more specifically by informing us about the installation of a VO2 dependence, and therefore of an anaerobic metabolism. Patients are randomized in 2 groups : Control group: hemodynamic management of patients is done according to usual practices by maintenance of blood pressure by norepinephrine as well as optimization of Systolic Voume (SV) by vascular filling and use of dobutamine if necessary. Experimental group: perioperative hemodynamic management is based on an algorithm that includes RQ measurement and includes volume expansion, norepinephrine, FiO2 enhancement, RBC transfusion and dobutamine. Primary and secondary outcomes are recorded 1,2,7 and 30 days after the surgery.

DETAILED DESCRIPTION:
• Background : The measurement of the inspired / expired fractions in O2 and CO2 is part of the daily monitoring of the intubated-ventilated patient in the operating theater. Changes in EtCO2 may reflect changes in metabolic CO2 production (VCO2), and oxygen extraction from the body (SvO2). The inspired / exhaled oxygen difference is an indirect reflection of the oxygen consumption (VO2). The ratio of VCO2 to VO2 (respiratory quotient (RQ)) is a non-invasive indirect measure of anaerobic metabolism of the patient, and an indirect reflection of tissue perfusion.

Some studies, including a recent one carried out by our center, showed that the RQ was linked to the appearance of anaerobic metabolism and to the postoperative evolution of the patient. The RQ was correlated with arterial lactate levels and predicted the occurrence of postoperative complications. Thus, the RQ can be a reliable, continuous, non-invasive marker of anaerobic metabolism in the operating room and therefore of the adequacy of arterial oxygen Transport (TaO2) with respect to the VO2 of the patient

* Purpose : Th investigators hypothesize that a hemodynamic optimization in major surgery individualized by non-invasive continuous measurement of the RQ would optimize TaO2 more specifically by informing us about the installation of a VO2 dependence, and therefore of an anaerobic metabolism.
* Brief summary:

The measurement of the inspired / expired fractions in O2 and CO2 is part of the daily monitoring of the intubated-ventilated patient in the operating theater. The ratio of VCO2 to VO2 (respiratory quotient (RQ)) is a non-invasive indirect measure of anaerobic metabolism of the patient, and an indirect reflection of tissue perfusion. We hypothesize that a hemodynamic optimization in major surgery individualized by non-invasive continuous measurement of the RQ would optimize TaO2 more specifically by informing us about the installation of a VO2 dependence, and therefore of an anaerobic metabolism. Patients are randomized in 2 groups : Control group: hemodynamic management of patients is done according to usual practices by maintenance of blood pressure by norepinephrine as well as optimization of Systolic Voume (SV) by vascular filling and use of dobutamine if necessary. Experimental group: perioperative hemodynamic management is based on an algorithm that includes RQ measurement and includes volume expansion, norepinephrine, FiO2 enhancement, RBC transfusion and dobutamine. Primary and secondary outcomes are recorded 1,2,7 and 30 days after the surgery.

Number of groups and description of groups :

2 groups Control group: hemodynamic management of patients is done according to usual practices by maintenance of blood pressure by norepinephrine as well as optimization of SV by vascular filling and use of dobutamine if necessary.

Experimental group: perioperative hemodynamic management is based on an algorithm that includes RQ measurement and includes volume expansion, norepinephrine, FiO2 enhancement, RBC transfusion and dobutamine.

• Interventions : Control group: hemodynamic management of patients is done according to usual practices by maintenance of blood pressure by norepinephrine as well as optimization of SV by vascular filling and use of dobutamine if necessary.

Experimental group: perioperative hemodynamic management is based on an algorithm that includes RQ measurement and includes volume expansion, norepinephrine, FiO2 enhancement, RBC transfusion and dobutamine.

The primary outcome is defined by at least one organ failure within 7 days postoperatively.

The duration of participation of each patient is 30 days and total research term is 49 months

* Number of subjects : 350
* Statistical analysis : The null hypothesis will be rejected in favor of the alternative hypothesis (there is a difference) using a test of χ2 or a Fisher test according to the frequency of the complications with a risk of the first bilateral species of 5%.
* Key-words : respiratory quotient, post opérative complications, anaerobic metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal, orthopedic or vascular surgery with general anesthesia
* ASA score ≥ II
* Estimated duration of surgery> 2 hours
* Consent signed.
* Affiliation to a social security scheme

Exclusion Criteria:

* Untreated or unbalanced severe hypertension under treatment.
* Preoperative renal failure dialyzed.
* Acute heart failure.
* Acute coronary insufficiency.
* Vascular surgery with kidney plasty.
* Cardiac surgery.
* Permanent laparoscopy.
* Preoperative shock state.
* Refusal of patient's participation
* Pregnant woman, parturient or breastfeeding.
* Patient under guardianship or trusteeship, under the protection of justice or private public law.
* Anesthesia with loco-regional anesthesia (spinal anesthesia and epidural).
* Acute respiratory distress syndrome (PaO2 / FiO2 ratio <300).
* Chronic Respiratory Failure with Home Oxygen Therapy.
* Patient already included in another therapeutic trial with an experimental molecule.
* Emergency anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
organ failure | 7 days postoperatively
  at least one organ failure within 7 days postoperatively. • Organ failure is defined according to the recommendations of the European Anesthesia Society (ESA) and the European Resuscitation Society (ESICM).
mortality rate at day 30 | 30 days

SECONDARY OUTCOMES:
the length of stay in the hospital | 30 days
the SOFA score at day1 | 1 day
  The sequential organ failure assessment score (SOFA score), previously known as the sepsis-related organ failure assessment score, is used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The SOFA scoring system is useful in predicting the clinical outcomes of critically ill patients.According to an observational study at an Intensive Care Unit (ICU) in Belgium, the mortality rate is at least 50% when the score is increased, regardless of initial score, in the first 96 hours of admission, 27% to 35% if the score remains unchanged, and less than 27% if the score is reduced. Score ranges from 0 (best) to 24 (worst) points.
the SOFA score at day2 | 2 days
  The sequential organ failure assessment score (SOFA score), previously known as the sepsis-related organ failure assessment score, is used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The SOFA scoring system is useful in predicting the clinical outcomes of critically ill patients.According to an observational study at an Intensive Care Unit (ICU) in Belgium, the mortality rate is at least 50% when the score is increased, regardless of initial score, in the first 96 hours of admission, 27% to 35% if the score remains unchanged, and less than 27% if the score is reduced. Score ranges from 0 (best) to 24 (worst) points.
the SOFA score at day7 | 7 days
  The sequential organ failure assessment score (SOFA score), previously known as the sepsis-related organ failure assessment score, is used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The SOFA scoring system is useful in predicting the clinical outcomes of critically ill patients.According to an observational study at an Intensive Care Unit (ICU) in Belgium, the mortality rate is at least 50% when the score is increased, regardless of initial score, in the first 96 hours of admission, 27% to 35% if the score remains unchanged, and less than 27% if the score is reduced. Score ranges from 0 (best) to 24 (worst) points.
total volume of fluid intraoperatively | 30 days
Plasma creatinine measured on day 0, day 1, day 2 and day 7 postoperatively | 7 days
Plasma lactate measured on day 1, day 2 and day 7 postoperatively | 7 days
C Reactive protein measured on day1, day2 and day7 postoperative | 7 days
Troponin Tc measured on day1, day2 and day7 postoperatively | 7 days
(NT pro) Brain Natriuretic Peptide ((NT pro) BNP) measured at day1, day2 and day7 postoperative | 7 days
the incidence of each complication | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Bar, Dr, Principal Investigator — CHU Amiens
Locations (1):
- BAR, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bar S, Boivin P, El Amine Y, Descamps R, Moussa M, Abou Arab O, Fischer MO, Dupont H, Lorne E, Guinot PG. Individualized hemodynamic optimization guided by indirect measurement of the respiratory exchange ratio in major surgery: study protocol for a randomized controlled trial (the OPHIQUE study). Trials. 2020 Nov 23;21(1):958. doi: 10.1186/s13063-020-04879-x. PMID 33228773
- [Result] Bar S, Moussa MD, Descamps R, El Amine Y, Bouhemad B, Fischer MO, Lorne E, Dupont H, Diouf M, Guinot PG; OPHIQUE study group. Determinants of postoperative complications in high-risk noncardiac surgery patients optimized with hemodynamic treatment strategies: A post-hoc analysis of a randomized multicenter clinical trial. J Clin Anesth. 2024 May;93:111325. doi: 10.1016/j.jclinane.2023.111325. Epub 2023 Nov 22. PMID 37992534
- [Result] Bar S, Moussa MD, Descamps R, El Amine Y, Bouhemad B, Fischer MO, Lorne E, Dupont H, Diouf M, Guinot PG; OPtimization Hemodynamic Individualized using the respiratiory QUotiEnt (OPHIQUE) Trial Group. Respiratory Exchange Ratio guided management in high-risk noncardiac surgery: The OPHIQUE multicentre randomised controlled trial. Anaesth Crit Care Pain Med. 2023 Aug;42(4):101221. doi: 10.1016/j.accpm.2023.101221. Epub 2023 Mar 21. PMID 36958473